CLINICAL TRIAL: NCT02261168
Title: Day-night Rhythm in Human Skeletal Muscle Metabolism
Brief Title: Day-Night Rhythm in Human Skeletal Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METC143027; NL49363.068.14 (Registry Identifier: Toetsing Online)
Record Dates: First submitted 2014-09-24; First posted 2014-10-10 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Mellitus, Type 2; Insulin Resistance
Keywords: Circadian Rhythm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Standardized living protocol (Other): Subjects are kept at the research facility to adhere to a standardized living protocol, mimicking a normal daily living situation. During the study, multiple tests will be performed, including muscle biopsies, blood draws, MRS measurements and indirect calorimetry.
  Interventions: Other: Standardized living protocol

INTERVENTIONS:
Other: Standardized living protocol — Subjects stay at the research facility for 44 hours and adhere to a standard sleeping, eating and activity protocol. During this protocol, multiple measurements will be performed including skeletal muscle biopsies (m. vastus lateralis), blood draws, indirect calorimetry and MRS measurements.

SUMMARY:
This study evaluates the existence of a day-night rhythm in skeletal muscle energy metabolism in healthy lean subjects. Subjects will stay at the research facility for 44 hours with a standardized living protocol during which several measurements of skeletal muscle and whole body energy metabolism will be performed.

DETAILED DESCRIPTION:
Recent evidence from both observational and experimental studies indicates that disobeying our normal day-night rhythm negatively influences our metabolic and cardiovascular health, possibly leading to obesity and type 2 diabetes mellitus (T2DM). An important hallmark of obesity and T2DM is a decreased skeletal muscle mitochondrial function. Interestingly, recent research indicates that also skeletal muscle mitochondrial function under the influence of a day-night rhythm. The main objective of this study is to investigate the presence of a day-night rhythm in skeletal muscle energy metabolism (in particular mitochondrial function) of healthy young participants. Therefore, subjects will stay at the research unit for 44 hours, with standardized meals and sleeping time. During this period we will take five muscle biopsies, perform indirect calorimetry measurements and blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Healthy (as determined by dependent physician based on medical questionnaire)
* Male
* Age: 18-35 years
* Normal BMI (18-25 kg/m2)
* Regular sleeping time (normally 7-9h daily)

Exclusion Criteria:

* Extreme early bird or extreme night person (score ≤30 or ≥70 on MEQ-SA questionnaire)
* Heavily varying sleep-wake rhythm
* Shiftwork during last 3 months
* Travel across >1 time zone in the last 3 months
* Engagement in exercise > 2 hours total per week
* Using >400mg caffeine daily
* Smoking
* Unstable body weight (weight gain or loss > 3kg in the last 3 months)
* Significant food allergies/intolerance (seriously hampering study meals)
* Participation in another biomedical study within 1 month before the first study visit
* Any contra-indication to Magnetic Resonance Imaging (MRI) scanning

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Day-night rhythm in skeletal muscle mitochondrial respiration | 40 hours.
  O2-flux (pmol/mg/s) measured with high resolution respirometry upon administration of different substrates

SECONDARY OUTCOMES:
Day-night rhythm in whole-body energy metabolism | 40 hours.
  Energy expenditure (kJ/min), glucose oxidation (g/min) and fat oxidation (g/min) measured by indirect calorimetry
Day-night rhythm in muscle DNA, mRNA and protein levels of markers involved in molecular clock and mitochondrial metabolism. | 40 hours.
  Quantify mRNA and protein levels by qPCR or micro-array and Western blots
Day-night rhythm of in markers of normal day-night rhythm (cortisol, melatonin, core body temperature) | measured during the 2nd study day
  Blood cortisol and melatonin levels and core body temperature measured by an ingested telemetric pill.
Day-night rhythm in blood metabolic compounds (e.g. glucose, insulin, FFA's, cholesterol) | measured during the 2nd study day
Day-night rhythm of molecular clock mRNA and protein levels in blood PBMC's | measured during the 2nd study day
  Measured by qPCR and Western Blots
Change in liver volume and liver lipid concentration during the day | First study day 6 PM, second study day 7 AM
  Measured by Magnetic Resonance Imaging and -Spectroscopy (MRI/MRS). Lipid signals in the MRS spectra will be quantified while suppressing the strong water signal in the region of interest (right liver lobe)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, PhD, Principal Investigator — Professor
Locations (1):
- Maastricht University, Maastricht, Netherlands